CLINICAL TRIAL: NCT06047301
Title: Pathways, a Hope-Based Intervention to Support Personal Goal Pursuit, Mental Health, and Quality of Life During Treatment for Advanced Lung Cancer
Brief Title: Pathways, a Hope Intervention to Support Personal Goal Pursuit, Mental Health, and Quality of Life During Advanced Lung Cancer Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laurie McLouth (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Laurie McLouth, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 87901; 1R01CA283929-01 (NIH)
Record Dates: First submitted 2023-09-14; First posted 2023-09-21 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Lung Cancer
Keywords: advanced cancer; palliative; supportive oncology; psychosocial intervention
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pathways (Experimental): Pathways focuses on increasing patient hope to support personal goal pursuit during treatment for advanced lung cancer.
  Interventions: Behavioral: Pathways
- Enhanced Usual Care (Active Comparator): Enhanced Usual Care focuses on providing patients with education around common lung cancer concerns (e.g., pain and fatigue management) and resources to support them (e.g., supportive services available nationally and at the treating cancer center).
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Pathways — Delivered by a nurse or other healthcare provider, includes 2 in-person sessions, and phone check-ins, and occurs primarily during infusion visits. Includes a Pathways Toolkit with handouts on values and goal setting, as well as resources on symptom management, lung cancer stigma, communication strategies, and other cancer center resources.
  Arms: Pathways
Behavioral: Enhanced Usual Care — Pathways Toolkit handouts on symptom management, lung cancer stigma, communication strategies, and other cancer center resources provided to participants. The Toolkit will be reviewed with patients in person to orient them to its purpose and contents.
  Arms: Enhanced Usual Care

SUMMARY:
This study will compare the effects of a brief supportive intervention, called Pathways, against enhanced usual care on the mental health and quality of life of people undergoing treatment for advanced lung cancer. Patients will complete baseline survey measures and be randomized to intervention. Survey measures will be collected again mid-intervention, post-intervention and at 6- and 12-week follow-up, with analyses focused on changes pre- to post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* New or recurrent AJCC 8th edition stage 3b, 3c, or IV non-small cell lung cancer, extensive stage small cell lung cancer
* 18 years of age or older
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2/Karnofsky 60-100
* 3-12 weeks into systemic, infusion-based treatment (chemotherapy, immunotherapy, chemo-immunotherapy)
* Past month distress score (per electronic health record) of 3/10 or higher OR a Rotterdam Symptom item score of 2 or higher for psychological distress items.

Exclusion Criteria:

* Unstable brain metastases (i.e., progressive neurological deficits, inadequately controlled seizures, or requiring escalated steroid doses)
* Cognitive (i.e., dementia) or psychiatric condition (e.g., psychotic disorder) for which participating would be inappropriate
* Receiving overlapping palliative care or psychological services at the cancer center
* Unable to speak and read English.
* Hearing or visual impairment that precludes study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2023-11-29 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in PROMIS Depression Short Form Scores | 12 weeks (Baseline, Post-Intervention)
  Depression symptoms will be measured using the PROMIS Depression Short Form 6a: 6 items are responded to on a scale of 1 = never to 5 = always. Raw scores range from 6 to 30.
  Higher scores indicate more depression.
Change in State Hope scores | 12 weeks (Baseline, Post-Intervention)
  Hope will be measured using Snyder's State Hope Scale. 6 items responded to on a scale of 1 = definitely false to 8 = definitely true. Raw scores range from 6 to 48. Items are summed for a total score. Higher scores indicate higher hope.

SECONDARY OUTCOMES:
Change in PROMIS Anxiety Short Form Scores | 12 weeks (Baseline, Post-Intervention)
  Anxiety symptoms are measured using the PROMIS Anxiety Short Form 4a. 4 items are responded to on a scale of 1 = never to 5 = always. Raw scores range from 4 to 20. Higher scores indicate more anxiety.
Change in Demoralization Scale II Scores | 12 weeks (Baseline, Post-Intervention)
  Demoralization symptoms are measured using the Demoralization Scale II: 16 items are responded to on a scale of 0 = never to 2 = always; Raw scores range from 0-32. Higher scores indicate more demoralization.
Change in PROMIS 15a positive affect scores | 12 weeks (Baseline, Post-Intervention)
  Positive affect is measured using the PROMIS 15a positive affect form. Higher scores indicate more positive affect. Items are responded to on a scale of 1 = never to 5 = always. Raw scores range from 15 to 45. Higher scores indicate more positive affect.
Change in FACIT-Spiritual Well-being Meaning/Peace Subscale Scores | 12 weeks (Baseline, Post-Intervention)
  Meaning/Peace is measured using the FACIT-Spiritual Well-being Meaning/Peace Subscale. 8 items are responded to on a scale of 0 = not at all to 4 = very much. Raw scores range from 0-32. Higher scores indicate more meaning/peace.
Change in FACT-G7 Quality of Life Scores | 12 weeks (Baseline, Post-Intervention)
  Quality of Life is measured using the FACT-G7. 7 items are responded to on a scale of 0 = not at all to 4 = very much to assess physical, emotional, and functional wellbeing. Raw scores range from 0 to 28. Higher scores indicate better quality of life.
Change in PROMIS Satisfaction with Participation in Social Roles 8a Short Form Scores | 12 weeks (Baseline, Post-Intervention)
  Satisfaction with Social Activities and Roles is measured using the ROMIS Satisfaction with Participation in Social Roles 8a Short Form. 8 items are responded to on a scale of 1 = not at all to 5 = very much. Raw scores range from 8 to 40. Higher scores indicate better function.

CONTACTS AND LOCATIONS:
Overall Officials: Laurie McLouth, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
Data Description: The proposed research will include clinical and patient-reported outcome data from approximately 234 participants with advanced stage lung cancer. Patients will complete surveys prior to randomization, mid-intervention period, post-intervention, and at follow-ups. In addition to these survey data, disease and medical treatment information will be abstracted from the electronic health record, including cancer treatments received, performance status, hospitalizations, and death.
  Data Archive: Data from this study will be submitted to ICPSR (Inter-university Consortium for Political and Social Research), which will make de-identified data available as described under "access criteria."
Supporting Information: Study Protocol, ICF
Time Frame: Data will be submitted to ICPSR a year after study completion. ICPSR will archive the full dataset and its documentation for the long term.
Access Criteria: ICPSR will make the data available to the broader research community. Files for public use (direct and indirect identifiers removed) will be accessible directly through the ICPSR website. After agreeing to Terms of Use, users with an ICPSR MyData account and an authorized IP address from a member institution may download the data, and non-members may purchase the files.